CLINICAL TRIAL: NCT06267105
Title: Clinical Study to Compare Functional Results in Patients Affected by Trigger Finger When Surgery is Performed Through a Transverse or Longitudinal Surgical Incision in the Skin.
Brief Title: A Clinical Study to Compare Functional Outcomes After Surgery Using a Transverse or Longitudinal Surgical Incision in the Skin.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Corona Poy, Doctor, Corporacion Parc Tauli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A1-LORT
Record Dates: First submitted 2024-01-31; First posted 2024-02-20 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Functional Disturbance as Result

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longitudinal incision (Experimental): Incision performed longitudinally
  Interventions: Procedure: Longitudinal incision
- Transverse incision (Experimental): Incision performed transversally
  Interventions: Procedure: Transverse incision

INTERVENTIONS:
Procedure: Longitudinal incision — Incision performed longitudinally
  Arms: Longitudinal incision
Procedure: Transverse incision — Incision performed transversally
  Arms: Transverse incision

SUMMARY:
Trigger finger is a common pathology in the hand. Patients suffer from pain and depending on which tasks, patients have difficulty to perform them. Its treatment in initial and less serious phases includes conservative measures, but failure of these may require releasing the trigger finger with surgery. The surgical technique performed for trigger finger is the opening of the A1 pulley, the skin incisions used for this surgery are various (transverse, longitudinal, oblique). Trigger finger surgery presents good results in terms of resolution, but complications may also occur. The reason for this study is to assess whether there are functional differences using the Dash scale when we perform a transverse or longitudinal incision in trigger finger surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age.
* Clinical diagnosis of trigger finger grade II to IV.

Grade I (pre-trigger) Pain, history of entrapment, but not demonstrable on physical examination, tenderness over the A1 pulley.

Grade II (active) Demonstrable entrapment, but the patient can actively extend the finger.

Grade III (passive) Demonstrable entrapment, patient requires passive extension IIIA or inability to actively flex IIIB.

Grade IV (contracture) Demonstrable entrapment with fixed flexion contracture of the PIP.

Exclusion Criteria:

* Thumb
* Polydigital
* Allergy to local anesthetics and/or vasoconstrictor agents.
* Previous surgery
* Patients who, in the researcher's opinion, are not good candidates for the study (e.g. inability to comply with the follow-up program, comorbidity, poor physical or mental health in general, drug or alcohol abuse problems...).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Functional improvement of the patient after surgery | Immediately after surgery
  functional improvement of the patient after surgery, which will be assessed with the Dash scale, 1 being difficult while 5 being unable

SECONDARY OUTCOMES:
Surgeon comfort | Immediately after surgery
  Ecellent, good, poor
Resolution | 1, 3 and 6 months
  Presence or absence of engagment
Flushed | 1, 3 and 6 months
  Red or not red
Pain feeling | 1, 3 and 6 months
  EVA scale from 0 to 10, being 10 a lot of pain
Contracture | 1, 3 and 6 months
  Range of motion in degrees
Infection | 1, 3 and 6 months
  Septic signs such the area is red, hot, swelling or has drain pus
Nerve injury | 1, 3 and 6 months
  Allen test to evaluate correct circulation, the hand should turn white when pressing
Return to work | 1, 3 and 6 months
  How many weeks after surgery
Reincorporation to activities | 1, 3 and 6 months
  How many weeks after surgery
Sensitivity Test | 1, 3 and 6 months
  In a scale from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Parc taulí, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mohd Rashid MZ, Sapuan J, Abdullah S. A randomized controlled trial of trigger finger release under digital anesthesia with (WALANT) and without adrenaline. J Orthop Surg (Hong Kong). 2019 Jan-Apr;27(1):2309499019833002. doi: 10.1177/2309499019833002. PMID 30852960
- [Background] Kazmers NH, Holt D, Tyser AR, Wang A, Hutchinson DT. A prospective, randomized clinical trial of transverse versus longitudinal incisions for trigger finger release. J Hand Surg Eur Vol. 2019 Oct;44(8):810-815. doi: 10.1177/1753193419859375. Epub 2019 Jul 4. PMID 31272265
- [Background] Kloeters O, Ulrich DJ, Bloemsma G, van Houdt CI. Comparison of three different incision techniques in A1 pulley release on scar tissue formation and postoperative rehabilitation. Arch Orthop Trauma Surg. 2016 May;136(5):731-7. doi: 10.1007/s00402-016-2430-z. Epub 2016 Feb 29. PMID 26926477